CLINICAL TRIAL: NCT02028299
Title: Estimation of Pulmonary Vascular Resistance by Contrast Echocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 060922
Record Dates: First submitted 2013-08-20; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Pulmonary Vascular Resistance; Right Heart Catheterization
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2D doppler echo with Definity solution (Experimental): Study subjects will already be scheduled for right heart catheterization to diagnose pulmonary hypertension. Prior to the catheterization, each subject will have a 2D doppler echocardiogram with Definity solution as well.
  Interventions: Procedure: 2D doppler echo with Definity solution

INTERVENTIONS:
Procedure: 2D doppler echo with Definity solution — Correlate right heart catheterization results with results from 2D doppler echo with Definity Solution
  Other Names: Definity solution

SUMMARY:
An echocardiogram using Definity contrast can provide the same information as the standard right heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergo right heart catheterization at the George Washington University Hospital

Exclusion Criteria:

* Patients with known or suspected right-to-left bi-directional or transient right-to-left shunts or pulmonary arteriovenous malformations, previously documented moderate to severe tricuspid regurgitation or moderate to severe pulmonary regurgitation, evidence of right ventricular hypokinesis, or prior adverse reaction to Definity or hypersensitivity to perflutren

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Measure Pulmonary Vascular Resistance using 2D Doppler Echocardiogram w/Definity Solution | Two Years
  Correlation coefficients between the technique above the the gold standard right heart catheterization measures of pulmonary vascular resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Choi, MD, Principal Investigator — Medical Faculty Associates, Inc.